CLINICAL TRIAL: NCT01286389
Title: Caloric Restriction in Obese Patients With Mild Cognitive Impairment: Effects on Adiposity, Comorbidity and Cognition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Nídia Celeste Horie, MD, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0706/10 CAPPesq
Record Dates: First submitted 2011-01-27; First posted 2011-01-31 (Estimated); Last update posted 2014-11-05 (Estimated); Status verified 2014-11

CONDITIONS: Mild Cognitive Impairment; Obesity
Keywords: Mild cognitive impairment; Dementia; Obesity; Overweight; diet; caloric restriction; body composition; weight loss
MeSH Terms: conditions — Cognitive Dysfunction; Obesity; Dementia; Overweight; Weight Loss | interventions — Caloric Restriction; Diet

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional medical care (Active Comparator): Conventional medical care, geriatric consultations at least 6 times in 12 months, short lifestyle counseling (exercise+healthy diet)
  Interventions: Other: medical care
- caloric restriction +medical care (Experimental): Nutritional counseling individually and in groups, aiming to promote weight loss (10% of body weight) through caloric restriction, +Conventional medical care, geriatric consultations at least 6 times in 12 months, short lifestyle counseling (exercise)
  Interventions: Other: medical care; Behavioral: caloric restriction

INTERVENTIONS:
Other: medical care — Conventional medical care, geriatric consultations at least 6 times in 12 months, short lifestyle counseling (exercise+healthy diet)
Behavioral: caloric restriction — Nutritional guidance: through at least 2 individual assistance and group sessions, lasting 1 hour, weekly for 4 months, and biweekly for 2 months and monthly thereafter (26-28 meetings/1year).The diet plan will recommend a deficit from 500 to 750 kcal/day in order to promote loss of about 0.5kg/week, containing 1g/kg of protein per day (minimum 1200kcal/day), high in fiber, vegetables and whole foods. The goal of weight loss will be 10% of initial weight. Group activities consist of lectures on nutrition education, food composition and its importance to health, food preparation techniques, self-monitoring weight, eating behavior and count calories.
  Other Names: diet
  Arms: caloric restriction +medical care

SUMMARY:
Obesity has been associated with cognitive impairments, lower blood flow, metabolic activity and brain volume. Obesity in adulthood is a risk factor for Alzheimer's disease in the elderly. The mild cognitive impairment (MCI) is a condition that may precede dementia. We hypothesized that promotion of weight loss in obese people with MCI, through caloric restriction could lead to improvement in cognitive performance or reduction in the rate of decline and decreased risk of dementia. A sample of 80 patients aged ≥ 60 years, obese, with MCI, will be randomized to two groups that will be followed for 12 months. The control group will receive conventional medical care. The intervention group will receive nutritional counseling individually and in groups, aiming to promote weight loss through caloric restriction, and medical monitoring. Before and after intervention patients will be evaluated for anthropometry, body composition, physical performance, control of comorbidities, laboratory tests (glucose, insulin, lipid profile, leptin, adiponectin, interleukin 6, tumor necrosis factor alpha, CRP), Genotyping apolipoprotein E, neuropsychological battery, questionnaires about activities of daily living, physical activity and diet.

DETAILED DESCRIPTION:
Objectives: To evaluate the cognitive performance of obese patients with MCI and the effect of weight loss induced by caloric restriction on cognition, conversion to dementia, to assess weight loss, changes in inflammatory and metabolic parameters, change in physical capacity, performance in neuropsychological tests and correlate with effects of the intervention. Methods: The patients will be randomized to two groups that will be followed for 12 months. The control group will receive conventional medical care. The intervention group will receive nutritional counseling individually and in groups, aiming to promote weight loss (10% of body weight) through caloric restriction, and medical monitoring. Everyone will be advised to physical activity. Before and after 12 months patients will be evaluated for anthropometry, body composition, physical performance, control of comorbidities, laboratory tests (glucose, insulin, lipid profile, leptin, adiponectin, interleukin 6, tumor necrosis factor alpha, CRP), Genotyping apolipoprotein E, neuropsychological battery, questionnaires about activities of daily living, physical activity and diet.

ELIGIBILITY:
Inclusion Criteria:

* body mass index (BMI) ≥ 30 kg/m2
* independent for most of the instrumental activities of daily life;
* literate;
* able to walk,
* diagnosis of mild cognitive impairment

Exclusion Criteria:

* weight loss greater than 3 kg over the past two months,
* presence of uncontrolled disease that potentially interfere with metabolism and weight gain or whose treatment would influence the cognitive performance, such as major depression, bulimia, hypothyroidism, Cushing's disease, heart failure, neoplasia in the last 3 years, alcoholism, infectious diseases and auto-immune activity;
* use of anti-obesity drugs, benzodiazepines, neuroleptics or estrogen replacement therapy in the past 2 months;
* previous bariatric surgery,
* severe sensory deficit

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2011-01; Primary Completion 2013-05 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Neuropsychological test performance | baseline and 12 months
  Montreal Cognitive Assessment (MoCA), Mini Mental State Examination (MMSE), Subjective Memory Complaints scale and CAMcog from CAMDEX (The Cambridge Examination for Mental Disorders of the Elderly, The Rivermead Behavioural Memory, The Wisconsin Card Sorting Task, trail making test part A and B, The Rey auditory-verbal learning test, semantic and phonologic verbal fluency test, digits (WAIS-III), vocabulary (WAIS - III), matrix (WAIS - III)
Diagnosis of dementia | 12 months
  The diagnosis of dementia will be given from the DSM IV TR: The diagnosis of Alzheimer's disease will be defined according to DSM IV.
Weight loss | 12 months
  anthropometry (weight, height, BMI, waist circumference, hip circumference), body composition by bioimpedance

SECONDARY OUTCOMES:
plasma biomarkers | 0 and 12 months
  glucose, insulin, lipid profile, leptin, adiponectin, interleukin 6, tumor necrosis factor alpha, CRP
Genotyping apolipoprotein E | baseline
  The genotype is a covariate to assess response to treatment
Charlson comorbidity index | 0 and 12 moths
International physical activity questionnaire- short version (IPAQ) | 0 and 12 moths
Evaluation of Food Consumption | 0 and 12 moths
SPPB- Short physical performance battery | 0 and 12 moths
Blood pressure | 0 and 12 moths

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo Hapern, professor, Study Director — Sao Paulo University; Nídia Horie, Principal Investigator — pos graduation student of Sao Paulo University; Cintia Cercato, professor, Study Chair — Sao Paulo University
Locations (1):
- Hospital das Clínicas - Faculdade de Medicina da USP, São Paulo, São Paulo, Brazil